CLINICAL TRIAL: NCT02411162
Title: Skin Residency Study of Topically Applied GSK2894512 Cream in Healthy Volunteers
Brief Title: A Single Dose Phase I Exploratory Study in Healthy Volunteers With GSK2894512 Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201661
Record Dates: First submitted 2015-03-06; First posted 2015-04-08 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis; FLIM; chronic plaque psoriasis; healthy volunteers; GSK2894512; Skin residency
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Arm (Experimental): In Cohort 1, study medication (Cream A, 1%) will be applied as a thin layer onto a predefined area of the volar region of the forearm that is large enough to image and collect 3 biopsies (4 mm per biopsy). Vehicle will be applied on Day 1 only, onto a symmetrical location on the opposite forearm from Cream A. In cohort 2, subjects will be enrolled to evaluate Cream A (1%) and a different GSK2894512 Cream, Cream B (1%). Cream A, 1% and Cream B, 1% will be applied as a thin layer to the opposite forearms of the subject. Vehicle will be applied only on Day 1 to a separate area (at least 1.3 cm from study drug) of the forearm from where drug is applied. Both Cream A and Cream B will continue to be applied OD to the same area of the same forearm for 7 days.
  Interventions: Drug: Combination therapy GSK2894512 Cream A + GSK2894512 Cream B; Drug: Combination therapy Vehicle Cream A + Vehicle Cream B

INTERVENTIONS:
Drug: Combination therapy GSK2894512 Cream A + GSK2894512 Cream B — GSK2894512 Cream A, 1% (10mg/g) will be topically applied daily for 7 days as a thin layer onto an area of the volar region of one forearm (up to 1.5% body surface area) and GSK2894512 Cream B, 1% (10mg/g), will be topically applied daily for 7 days to the opposite forearm from Cream A, onto an area of the volar region of one forearm (up to 1.5% body surface area). Both the creams will be weighed to deliver approximately 3mg drug per 1cm^2 of skin.
Drug: Combination therapy Vehicle Cream A + Vehicle Cream B — Vehicle creams A and B will be supplied in individual tubes. Both the creams will be topically applied on Day 1 only to a separate area (at least 1.3 cm from study drug) of the forearm from where drug is applied.

SUMMARY:
This will be an open-label, non-randomized, single-center study to assess the residency of GSK2894512 in the skin of healthy adult male volunteers with normal barrier function. The study will have two parts, Cohort 1 (Part A) followed by Cohort 2 (Part B). The study will assess the residence time in human skin . The primary objective is to evaluate the residency time in skin following topical application of two formulations of GSK2894512 Cream. The total study duration will be of 15 days including 1 to 7 days of treatment period, 8 to 14 days of post treatment period and 1 day of follow up. The screening period will be up to 28 days prior to Baseline (Day 1).

ELIGIBILITY:
Inclusion Criteria:

* Males, between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Skin tone in the potential test site on the forearm such that erythema and other dermal reactions can be easily visualized, i.e. only Fitzpatrick skin types I (always burns; never tans), II (usually burns; tans with difficulty), III (sometimes mild burn; gradually tans), or IV (rarely burns; tans with ease) will be included. Determination of skin types is based on sunburn and tanning history in response to the first 30 to 45 minutes of sun exposure.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with values outside the normal range should always be excluded from enrolment.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Corrected QT interval (QTc) >450 milliseconds (msec)
* Concurrent conditions and history of diseases: Immunocompromized (eg, lymphoma, acquired immune deficiency syndrome (AIDS), Wiskott-Aldrich Syndrome or have a history of malignant disease within 5 years before the baseline visit, with the exception of basal and squamous cell cancers; Active acute bacterial, fungal or viral skin infection (e.g., herpes simplex, herpes zoster, chicken pox); Any other concomitant skin disorder (e.g., generalized erythroderma such as Netherton's Syndrome, atopic dermatitis or psoriasis), pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the test site evaluation or contraindicate participation; clinical signs of infection (viral, fungal or bacterial) within the treatment areas; other types of skin disease that may impact evaluation.
* Inability to evaluate the skin at and around the potential test sites on the forearms due to sunburn, unevenness in skin tones, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin damage or abnormality.
* Chronic or acute infection requiring treatment with systemic antibiotics, anti-virals, anti-parasitics, anti-protozoals, or anti-fungals within 4 weeks before the baseline visit, or superficial skin infections within 1 week before the screening visit.
* Planning a significant exposure to ultraviolet (UV) radiation (sun-bathing or tanning).
* Planning to use a sauna during the duration of the study or intending to swim more than once a week.
* Participation in a clinical drug or device research study within the previous 30 days.
* History of sensitivity to any of the study medications, local anesthesia, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Concomitant Medications: Investigational products and topical medications or products (including but not limited to self-tanning products, waxing products, benzoyl peroxide, salicylic acid, or sulphur) in the areas of testing.
* Contraindications: History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. . For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2015-09-24 (Actual); Study Completion 2015-09-24 (Actual)

PRIMARY OUTCOMES:
Residence time in skin following topical application of two formulations of GSK2894512 Cream | Up to Day 15
  Fluorescent lifetime imaging microscopy (FLIM) images will be evaluated to determine if GSK2894512 is detectable in skin. Drug concentrations can be quantified considering the: depth of penetration at each time point and the amount of fluorescence detected. Liquid Chromatography-Mass Spectrometry/Mass Spectrometry (LC-MS/MS) will also be used to measure the concentration of GSK2894512 from biopsies.

SECONDARY OUTCOMES:
Adverse events (AEs) monitoring after two formulations of GSK2894512 cream | Up to Day 15
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity, or; is a congenital anomaly/birth defect.
Composite of vital signs assessment including temperature, systolic and diastolic blood pressure and pulse rate of two formulations after two GSK2894512 cream | Up to Day 15
  Vital signs will be measured in semi-supine position after 5 minutes rest and will include temperature, systolic and diastolic blood pressure and pulse rate
Electrocardiogram (ECG) assessment after two formulations of GSK2894512 cream | Up to Day 15
  Single 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT interval for Bazett's formula (QTcB) intervals
Composite of abbreviated physical examination after two formulations of GSK2894512 cream | Up to Day 15
  Physical examination will include, at a minimum assessments of Cardiovascular, Respiratory, Gastrointestinal and Neurological systems. Height and weight will also be measured and recorded
Laboratory assessments after two formulations of GSK2894512 cream | Up to Day 15
  Laboratory assessments including haematology, clinical chemistry, and urinalysis
Local tolerability assessments after two formulations of GSK2894512 cream | Up to Day 15
  Tolerability will be evaluated on the basis of degree of local irritation.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Urbana, Illinois, United States

REFERENCES:
- See also: Results for study 201661 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201661?search=study&b'study_ids=201661'#rs